CLINICAL TRIAL: NCT02875574
Title: Improving the Management of Drug Resistant Tuberculosis in the UK
Acronym: UK_DR-TB
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/0074
Record Dates: First submitted 2016-07-25; First posted 2016-08-23 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Tuberculosis
Keywords: Isoniazid; Drug Resistance
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Drug: Any treatment regimen; Other: Bacterial mutation

INTERVENTIONS:
Drug: Any treatment regimen — Treatment regimen used to treat patient once isoniazid resistance known (exposure of interest for cohort study)
Other: Bacterial mutation — Resistance, compensatory or other mutation in the infecting strain of Mycobacterium tuberculosis (exposure of interest for nested case-control study)

SUMMARY:
The 'rising tide' of antimicrobial resistance is a source of concern across most infectious diseases. In the UK, for example, 6.8% of the ~8,500 tuberculosis patients seen in 2012 were resistant to the cheap and effective first-line drug isoniazid. It is of great importance to prevent the loss of current anti-tuberculosis drugs and preventing the spread of resistance by treating such patients as well as possible.

Currently, guidance on the best treatments for isoniazid resistant tuberculosis is inconsistent globally. Data from randomised controlled trials, the peak quality of evidence, is sparse. It is thus important that studies using pre-existing observational data are undertaken.

The investigators aim to use data and samples collected from Public Health England and National Health Service hospitals to determine a) the best treatments for patients with isoniazid resistant tuberculosis disease (cohort study) and b) how different causes of drug resistance in the infecting bacteria influence a) (nested case-control study). Eligible participants will have had isoniazid resistant tuberculosis (without associated rifampicin resistance) in England between 2009 and 2013 and will have been notified to Public Health England. The study will be conducted at University College London, National Health Service hospitals and Public Health England and will last until December 2017. Patient hospital records and disease surveillance records will be accessed and cultured bacteria from previously stored samples sequenced.

ELIGIBILITY:
Inclusion Criteria:

* Isoniazid resistant non-multidrug resistant tuberculosis patients.
* Notified to Public Health England's Enhanced Tuberculosis Surveillance System between 2009-2013.
* Adults aged 18 years and over.
* Patients not treated at private hospitals.

Exclusion Criteria:

* Non-notified patients.
* Individuals where the site of disease required more than 12 months of treatment.
* Individuals diagnosed post-mortem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with isoniazid resistant tuberculosis disease notified in England to Public Health England's Enhanced Tuberculosis Surveillance System 2009-13 who were not treated at private hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Treatment outcome | Up to 12 months after the start of treatment
  Negative versus positive treatment outcomes attributable to the treatment regimen commenced once isoniazid resistance known. Taken from clinical records.
  Also used to define cases and controls for nested case-control study.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS Foundation Trust, London, Greater London, United Kingdom